CLINICAL TRIAL: NCT00921115
Title: Combined Fulvestrant and Anastrozole as Neo-adjuvant Endocrine Therapy in Postmenopausal Women With Hormone Receptor Positive Invasive Breast Cancer
Brief Title: Anti-Hormone Therapy (With Anastrazole and Fulvestrant) Before Surgery to Treat Postmenopausal Women With Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11595; IRUSANAS0092 (Other: Astra Zeneca)
Record Dates: First submitted 2009-06-08; First posted 2009-06-16 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Invasive Breast Cancer
Keywords: hormone receptor positive; invasive breast cancer; endocrine therapy; Anastrazole; Fulvestrant; breast tumors; postmenopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arimidex + Faslodex (Experimental): Patients will have an Oncotype Dx performed and if the RS is <25, they will receive Anastrazole and Fulvestrant for 16 weeks.
  On day 28, subjects will be evaluated for side effects and a needle core biopsy (optional) will be obtained. Response evaluation will occur every 28 days. All treatment will continue for 4 months followed by breast surgery. After surgery, patients will be off study and will receive additional breast cancer therapy per their treating physician. Patients who develop progressive disease on protocol will be removed from the study and treated by their treating physician. The protocol will be closed after the last accrued patient has had surgery.
  Interventions: Drug: Fulvestrant; Drug: Anastrazole

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant IM on day 14 and on day 28 followed by day 28 of all subsequent cycles thereafter. Treatment will be continued for a total of 4 cycles.
  Other Names: Faslodex
Drug: Anastrazole — Anastrazole, 1mg by mouth every day of all 28 day cycles and continued for a total of 4 cycles
  Other Names: Arimidex

SUMMARY:
This study is being done to test the safety and effectiveness of two drugs, Anastrozole and Fulvestrant, used as combined therapy in the neo-adjuvant setting for hormone receptor positive invasive breast cancer.

DETAILED DESCRIPTION:
Hormonal therapies are generally preferred treatments of breast cancer because they have minimal side effects. Hormone receptor positive breast cancer generally does not respond very well to chemotherapy, which has many side effects. Hormonal therapy with a single drug such as Anastrozole is the main type of treatment used to reduce the risk of cancer recurrence. Whether a combination of Anastrazole nad Fulvestrant is effective and feasible is not known. This study is being done to answer this question.

This is a phase II single arm study. Patients will have an Oncotype Dx performed and only if the recurrence score is low or intermediate, they would be eligible. Eligible patients will receive Anastrazole and Fulvestrant for 16 week.

Subjects will receive Anastrazole 1 mg po q day and Fulvestrant 500 mg IM, day 1, day 14, day 28 and thereafter once every 28 days on outpatient basis. On day 28, subjects will be evaluated for side effects and clinically and a needle core biopsy (optional) will be obtained. If there is increase in Ki 67 by 50%, subjects will be taken off the study. Response evaluation will occur every 28 days during outpatient clinic visits. All treatment will continue until 4 months when patients will undergo surgical intervention. After surgery, patients will be off study and will receive additional breast cancer therapy at the discretion of their treating physician. Patients who develop progressive disease on protocol will be removed from the study and will then be treated at the discretion of the treating physician. The protocol will be closed after the last accrued patient has had surgery.

ELIGIBILITY:
Inclusion criteria

* Female patient > 18 years of age.
* Histologically proven invasive adenocarcinoma of the breast.
* Patients must be candidates for neoadjuvant treatment (Tumor size > 2cm and/or clinical N1 or N2).
* ER positive (> 10% of cells) and/or PgR positive (> 10% of the cells) and HER-2 negative disease (IHC 0 or 1+ and/or FISH negative, IHC 2+ and FISH negative)
* Menopausal status

  * Patients must be post-menopausal as defined by one of the following criteria:

    * Prior bilateral oophorectomy
    * 12 months since LMP with no prior hysterectomy
    * Patients > 55 years with prior hysterectomy
    * Patients < 55 years of age and with a prior hysterectomy without oophorectomy, estradiol and FSH levels must be consistent with the patient being postmenopausal.
  * Premenopausal or perimenopausal women who do not meet the postmenopausal criteria above are also eligible, but are required to undergo ovarian suppression with an LHRH agonist. Ovarian suppression can be initiated any time prior to or on day 1 of protocol therapy and must continue throughout protocol therapy.
* Performance status of 2 or better per SWOG criteria
* No prior chemotherapy or endocrine therapy for the current cancer diagnosis.
* If female of childbearing potential, pregnancy test is negative prior to initiation of ovarian suppression.
* Patients must be informed of the investigational nature of the study, and must sign an informed consent in accordance with the institutional rules.
* Oncotype Dx Recurrence Score </= 25.

Exclusion criteria

* Patients with metastatic disease.
* The presence of any other medical or psychiatric disorder that, in the opinion of the treating physician, would contraindicate the use of drugs in this protocol or place the subject at undue risk for treatment complications.
* Premenopausal without ovarian suppression.
* Pregnancy or lactation.
* Patients with concomitant or previous malignancies within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Patients with emotional limitations are excluded from study
* Platelets less than 100 x 109 /L
* Total bilirubin greater than 1.5 x ULRR
* ALT or AST greater than 2.5 x ULRR
* History of bleeding diathesis (i.e., disseminated intravascular coagulation [DIC], clotting factor deficiency) or long-term anticoagulant therapy (other than antiplatelet therapy).
* History of hypersensitivity to active or inactive excipients of fulvestrant (i.e. castor oil or Mannitol).
* Oncotype Dx Recurrence Score of >25.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qamar Khan, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arimidex + Faslodex: Patients will have an Oncotype Dx performed and if the RS is <25, they will receive Anastrazole and Fulvestrant for 16 weeks.
  On day 28, subjects will be evaluated for side effects and a needle core biopsy (optional) will be obtained. Response evaluation will occur every 28 days. All treatment will continue for 4 months followed by breast surgery. After surgery, patients will be off study and will receive additional breast cancer therapy per their treating physician. Patients who develop progressive disease on protocol will be removed from the study and treated by their treating physician. The protocol will be closed after the last accrued patient has had surgery.
  Fulvestrant: Fulvestrant IM on day 14 and on day 28 followed by day 28 of all subsequent cycles thereafter. Treatment will be continued for a total of 4 cycles.
  Anastrazole: Anastrazole, 1mg by mouth every day of all 28 day cycles and continued for a total of 4 cycles
Period: Overall Study
Arm/Group | Arimidex + Faslodex
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arimidex + Faslodex
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (PCR) Rate
Description: Pathologic complete response (PCR) rate with 4 months of neo-adjuvant combination endocrine therapy (Anastrazole and Fulvestrant).
Time Frame: 4 months
Population: Number of participants with PCR after 4 cycles of Neoadjuvant Endocrine Therapy
Measure: Number; unit: participants
Arm/Group | Arimidex + Faslodex
Number analyzed (Participants) | 42
participants | 0

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Arimidex + Faslodex
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 4/42
Other Adverse Events (participants affected / at risk) | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arimidex + Faslodex (N=42)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Valvular heart disease (Cardiac disorders) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arimidex + Faslodex (N=42)
Abdominal pain (Gastrointestinal disorders) | 1
Agitation (Psychiatric disorders) | 1
Allergic reaction (Immune system disorders) | 3
Anxiety (Psychiatric disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 9
Blurred vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Breast pain (Reproductive system and breast disorders) | 5
Bronchitis (Infections and infestations) | 1
Bruising (Skin and subcutaneous tissue disorders) | 1
standard error of the mean systolic ejection murmur (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Depression (Psychiatric disorders) | 5
change in hair texture (Skin and subcutaneous tissue disorders) | 1
actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 6
Dry eye syndrome (Eye disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Edema limbs (General disorders) | 3
worsening thyroid nodules requiring thyroidectomy (Endocrine disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 15
Fever (General disorders) | 3
Flashing vision (Eye disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gastric infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 4
Heartburn (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hot flashes (Endocrine disorders) | 21
Hypertension (Cardiac disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypotension (Cardiac disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
conjunctivitis (Infections and infestations) | 1
Infection, Upper airway NOS (Infections and infestations) | 1
Injection site reaction (Skin and subcutaneous tissue disorders) | 3
Insomnia (Psychiatric disorders) | 3
Joint pain (Musculoskeletal and connective tissue disorders) | 17
Joint-function (Musculoskeletal and connective tissue disorders) | 1 — decreased ROM 3/6 of bilateral upper extremities
Joint-function (Musculoskeletal and connective tissue disorders) | 1 — joint stiffness in the AM
Memory impairment (Nervous system disorders) | 1
Low Vitamin D (Metabolism and nutrition disorders) | 2
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (General disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 8
Pharyngitis (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Psychosis (Psychiatric disorders) | 1
upper airway congestion (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rhinitis infective (Infections and infestations) | 1
Rigors/chills (General disorders) | 3
Sinus tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1 — night sweats, hot flashes
Tinnitus (Ear and labyrinth disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1 — a piece of tooth broke off
Tremor (Nervous system disorders) | 1
Upper respiratory infection (Infections and infestations) | 2
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 3
Vaginal dryness (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Weight gain (Investigations) | 3
Weight loss (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No